CLINICAL TRIAL: NCT07030504
Title: The Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of SAL0133 Tablets in Chinese Adult Healthy Subjects
Brief Title: To Evaluate the Safety, Tolerability and Pharmacokinetic of SAL0133 Tablets in Chinese Adult Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL0133A101
Record Dates: First submitted 2025-06-10; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- SAD 50mg Fasting (Experimental): 6 subjects received active drug and 2 subjects received placebo once daily under fasting condition
  Interventions: Drug: SAL0133; Drug: SAL0133 placebo
- SAD 150mg Fasting (Experimental): 6 subjects received active drug and 2 subjects received placebo once daily under fasting condition
  Interventions: Drug: SAL0133; Drug: SAL0133 placebo
- SAD 300mg Fasting (Experimental): 6 subjects received active drug and 2 subjects received placebo once daily under fasting condition
  Interventions: Drug: SAL0133; Drug: SAL0133 placebo
- SAD 150mg Fed (Experimental): 6 subjects received active drug and 2 subjects received placebo once daily under fed condition
  Interventions: Drug: SAL0133; Drug: SAL0133 placebo
- SAD 300mg Fed (Experimental): 6 subjects received active drug and 2 subjects received placebo once daily under fed condition
  Interventions: Drug: SAL0133; Drug: SAL0133 placebo
- SAD 600mg Fed (Experimental): 6 subjects received active drug and 2 subjects received placebo once daily under fed condition
  Interventions: Drug: SAL0133; Drug: SAL0133 placebo
- MAD 150mg Fasting (Experimental): 6 subjects received active drug and 2 subjects received placebo once daily for seven days under fasting condition
  Interventions: Drug: SAL0133; Drug: SAL0133 placebo
- MAD 150mg Fed (Experimental): 6 subjects received active drug and 2 subjects received placebo once daily for seven days under fasting condition
  Interventions: Drug: SAL0133; Drug: SAL0133 placebo
- MAD 300mg Fed (Experimental): 6 subjects received active drug and 2 subjects received placebo once daily for seven days under fasting condition
  Interventions: Drug: SAL0133; Drug: SAL0133 placebo

INTERVENTIONS:
Drug: SAL0133 — once daily single dose or seven days multiple dose of SAL0133 tables
  Other Names: active drug group
Drug: SAL0133 placebo — once daily single dose or seven days multiple dose of SAL0133 placebo
  Other Names: placebo group

SUMMARY:
To evaluate the safety and tolerance of single and multiple administrations of SAL0133 tablets in adult healthy subjects in China receptivity.

DETAILED DESCRIPTION:
This study was divided into two parts: Part A and Part B. Part A was single-center, randomized, double-blind, and placebo control, single-dose escalation study (SAD) was conducted to evaluate the safety, tolerability and pharmacokinetic characteristics of SAL0133 tablets after a single dose. Furthermore, food effect would be preliminarily evaluated the influence of the pharmacokinetic characteristics of SAL0133 tablets in Part A. Part B was a single-center, randomized, double-blind, placebo controlled, multiple-dose escalation study was conducted to evaluate the safety, tolerability and pharmacokinetic characteristics of SAL0133 tablets after multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Participants have fully understood the trial's objectives, procedures, and potential adverse effects, and voluntarily signed informed consent form prior to the trial.
* Healthy male or female adults aged 18 to 65 years (inclusive).The gender ratio shall be no less than one third.
* Body weight ≥50 kg for male participants and ≥45 kg for female participants at screening, with a body mass index (BMI) between 19.0 and 26.0 kg/m2 (inclusive; BMI = body weight ÷ height2).
* No abnormalities or only slight abnormalities not clinically significant of tests/examinations (including physical examination, vital sign examination, blood routine, urine routine, blood biochemistry, coagulation function, five thyroid function tests, five pituitary function tests, serological virology, 12-lead electrocardiogram, normal chest position, abdominal B-ultrasound, etc) as judged by the investigator.
* The subject or their partner had no pregnancy plans during the study period and within one month after the last administration of the study drug, and the subjects do not donate sperm or eggs (oocytes, oocytes) for reproductive or assisted reproductive purposes.

Exclusion Criteria:

* Pregnant or lactating women, or women of child-bearing potential (WOCBP) with a positive pregnancy test at screening.
* A history of clinically significant drug allergies or allergic diseases (such as asthma, urticaria, eczema).
* Dermatitis, etc., or as determined by the investigator, it may or is clear to be effective against the research drug (including similar drugs and controls) or allergy to the medicine and any of its excipients. Clinically significant underlying liver diseases or medical history, including chronic hepatitis B, chronic hepatitis C, and alcohol liver disease and metabolism-related fatty liver disease, etc.
* Fever symptom or active infection within one week before the first administration of the drug.
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) and/or the total bilirubin (TBIL) is higher than the upper limit of the normal value (ULN) during screening.
* Have undergone gastric surgery, vagotomy, intestinal resection or any other procedures that might interfere with the gastrointestinal tract surgical procedures for peristalsis, pH or absorption.
* Have received active or attenuated vaccines within 4 weeks before screening. ·Any of the following drugs or treatments were used before the first administration.
* Drug or drug abuse, alcohol abuse, smoking addiction or special diet, etc. Any one of the antibody results is positive: Hepatitis B surface antigen, hepatitis C antibody, Treponema pallidum antibody, human immunodeficiency virus (HIV).
* Have participated in clinical studies of other drugs and taken any clinical study drugs within 3 months prior to the screening.
* Who have donated blood or lost ≥400 mL of blood, received blood transfusion or used blood products within 3 months prior to the screening.
* There is any disease history or current illness that may affect the safety of the subjects or the in vivo process of the investigational drug, including but not limited to the central nervous system, cardiovascular system, digestive system, respiratory system and endocrine system, urinary system, blood system, immune system, psychiatry, metabolic disorders, and those who have undergone gastrointestinal surgery (Except for cauditis surgery), etc.
* History of fainting from needles or blood, and it has been judged by the researcher to be of clinical significance.
* Any other reason, the researcher determines that the subject is not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The rate of AE | from Day 1 to Day 5 or Day 10
  The rate of AE occurred in the whole study
The rate of SAE | from Day 1 to Day 5 or Day 10
  The rate of SAE occurred in the whole study
blood pressure | from Day 1 to Day 5 or Day 10
  the change (mmHg) of blood pressure including SBP and DBP in the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Yang, M.D, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No